CLINICAL TRIAL: NCT06556134
Title: Oral Liposomal Iron Versus Injectable Iron Sucrose for Anemia Treatment in Non-Dialysis Chronic Kidney Disease Patients: A Non-Inferiority Study
Brief Title: Oral Liposomal Iron Versus Injectable Iron Sucrose for Anemia Treatment in Non-Dialysis Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Hassan II - Fès (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PREFER
Record Dates: First submitted 2024-08-10; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: hemoglobin; transferrin saturation; ferritin; liposomal iron; intravenous iron sucrose
MeSH Terms: interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP IV (Active Comparator): Group IV received intravenous iron-hydroxide sucrose complex (marketed as Fermed® 100mg), administered in a dose of 100 mg, diluted in 250 mL of normal saline, and infused weekly for a period of 3 month
  Interventions: Drug: Intravenous Iron Sucrose
- GROUP OS (Active Comparator): Group OS received one oral capsule per day, containing 30 mg of pyrophosphate liposomal iron and 70 mg of ascorbic acid (marketed as Lisofer® 30mg), for the same 3-month duration
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Intravenous Iron Sucrose — Intravenous iron-hydroxide sucrose complex administered in a dose of 100 mg, diluted in 250 mL of normal saline, and infused weekly for a period of 3 months
  Other Names: Fermed® 100mg
  Arms: GROUP IV
Drug: Oral Iron — One oral capsule per day, containing 30 mg of pyrophosphate liposomal iron and 70 mg of ascorbic acid
  Other Names: Lisofer® 30mg
  Arms: GROUP OS

SUMMARY:
This study aims to assess the comparative effects of intravenous and liposomal oral iron on hemoglobin levels in non-dialysis CKD patients. Additionally, it seeks to evaluate the rate of hemoglobin correction, iron reserve status during treatment, and therapeutic tolerance to these interventions.

DETAILED DESCRIPTION:
The last two and a half decades have seen erythropoiesis-stimulating agents (ESAs) and iron therapy at the forefront of managing anemia in chronic kidney disease (CKD) patients. While ESAs have demonstrated significant efficacy in alleviating anemia in this context, recent large-scale randomized controlled trials in both non-dialysis and dialysis CKD patients have shed light on their limitations. Attempts to normalize hemoglobin (Hb) levels with ESAs have shown no significant cardiovascular benefits but have been associated with increased risks of adverse events such as stroke and venous thromboembolism.

Consequently, there has been a reduction in ESA prescription and an increase in blood transfusions, coupled with a notable rise in the use of iron therapy due to its role in addressing hypo responsiveness to ESAs.

Anemia stands as a common complication in CKD, significantly impacting cardiovascular health and quality of life. While renal erythropoietin production deficit remains a primary cause, iron deficiency plays a pivotal role in CKD-related anemia genesis. Iron deficiency, whether absolute or functional, alongside an inflammatory block, often seen in CKD patients, accounts for the main reasons behind hypo responsiveness to erythropoiesis-stimulating agents.

The recent shift in focus from ESA-centered treatment to iron therapy has prompted debates regarding the ideal route of iron administration, particularly in non-dialysis CKD patients. Despite the benefits of oral iron-cost-effectiveness and ease of administration-its usage remains limited due to poor gastrointestinal absorption and high adverse event rates. Conversely, concerns about IV iron revolve around potential kidney damage, infections, atherosclerosis promotion, and other adverse reactions.

Given these considerations, our study aims to compare the efficacy of oral liposomal iron against IV iron in treating anemia in non-dialysis CKD patients in terms of :

1. Martial status under treatment.
2. Hemoglobin level and its correction speed.
3. Therapeutic tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study are age >18 years, eGFR ≤60 mL/min/1.73 m2 (Modification of Diet in Renal Disease equation: MDRD), Hb levels ≤12 g/dL, ferritin levels ≤100 ng/mL, transferrin saturation (TSAT) ≤25%, parathormone (PTH) serum levels between 30 and 300 pg/mL.

Exclusion Criteria:

* Exclusion criteria included presence of an inflammatory or infectious disease with a C-reactive protein (CRP) levels ≥6 mg/L at the beginning of the study ,surgical interventions in the last 3 months, hematological disorders including bleeding or blood transfusions in the last 6 months, malignancies, ongoing treatment with immunosuppressive drugs, severe malnutrition (BMI<20Kg/m² ; Albuminemia <32 g/L with normal values of C-reactive protein (CRP); Decrease in weight >5% in 1 month or >7.5% in 3 months), history of major CVD (Myocardial Infarction, Chronic Heart Failure, Stroke), chronic alcohol abuse, known hepatitis B or C infection, pregnant or lactating women, and need to start dialysis.

Withdrawal from the study occurs in the case of severe anemia needing an urgent blood transfusion or non-adherence and withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin elevation and its correction speed | Assessments were conducted at baseline (Month 0) and during all subsequent follow-up visits at months 1 (Month 1), 2 (Month 2), and 3 (Month 3), as well as the 2 months following the drug discontinuation (Month 4) and (Month 5)
  Clinical guidelines define a target hemoglobin range that indicates successful correction. Hemoglobin is measured in g/dL.

SECONDARY OUTCOMES:
Ferritin serum levels | Assessments of ferritin levels were conducted at baseline (Month 0) and during all subsequent follow-up visits at months 1 (Month 1), 2 (Month 2), and 3 (Month 3), as well as the 2 months following the drug discontinuation (Month 4) and (Month 5)
  Ferritin levels, measured in ng/mL, serve as a reliable indicator of the body's iron reserves, reflecting overall iron storage.
Transferrin saturation | Assessments of transferrin saturation were conducted at baseline (Month 0) and during all subsequent follow-up visits at months 1 (Month 1), 2 (Month 2), and 3 (Month 3), as well as the 2 months following the drug discontinuation (Month 4) and (Month 5)
  Transferrin saturation, expressed as a percentage (%), is a reliable indicator of iron availability in the body. The combination of ferritin levels (ng/mL) and transferrin saturation (%) provides the most reliable assessment of the body's iron status, offering a comprehensive view of both iron storage and availability.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Sqalli Houssaini, MD, Study Director — Laboratory of Epidemiology and Health Science Research, Sidi Mohammed Ben Abdellah University
Locations (1):
- Nephrology, Dialysis, and Transplantation, Hassan II University Hospital, Fes, Fès-Meknes, Morocco

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) often won't be shared with other researchers to protect participants' privacy and confidentiality. Sharing IPD could risk revealing personal information, even if anonymized, which might lead to re-identification. Additionally, there are ethical or legal obligations, informed consent restrictions, and concerns about misuse or misinterpretation of the data that necessitate keeping it restricted.

REFERENCES:
- [Result] Pisani A, Riccio E, Sabbatini M, Andreucci M, Del Rio A, Visciano B. Effect of oral liposomal iron versus intravenous iron for treatment of iron deficiency anaemia in CKD patients: a randomized trial. Nephrol Dial Transplant. 2015 Apr;30(4):645-52. doi: 10.1093/ndt/gfu357. Epub 2014 Nov 13. PMID 25395392
- [Result] Agrawal S, Sonawane S, Kumar S, Acharya S, Gaidhane SA, Wanjari A, Kabra R, Phate N, Ahuja A. Efficacy of Oral Versus Injectable Iron in Patients With Chronic Kidney Disease: A Two-Year Cross-Sectional Study Conducted at a Rural Teaching Hospital. Cureus. 2022 Jul 31;14(7):e27529. doi: 10.7759/cureus.27529. eCollection 2022 Jul. PMID 36060352
- [Result] Macdougall IC, Bock AH, Carrera F, Eckardt KU, Gaillard C, Van Wyck D, Roubert B, Nolen JG, Roger SD; FIND-CKD Study Investigators. FIND-CKD: a randomized trial of intravenous ferric carboxymaltose versus oral iron in patients with chronic kidney disease and iron deficiency anaemia. Nephrol Dial Transplant. 2014 Nov;29(11):2075-84. doi: 10.1093/ndt/gfu201. Epub 2014 Jun 2. PMID 24891437